CLINICAL TRIAL: NCT03297814
Title: A Randomized, Double Blind, Placebo Controlled Trial, Investigating the Effect of Intramuscular Injection of Allogenic Platelet Lysate for the Treatment of PAD
Brief Title: Use of Allogenic Platelet Lysate in Peripheral Arterial Disease (PAD)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sophia Al-Adwan (Other)
Responsible Party: Sponsor-Investigator, Sophia Al-Adwan, Clinical Co-ordinator, University of Jordan
Organization: University of Jordan (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PAD2UJCTC
Record Dates: First submitted 2017-08-08; First posted 2017-09-29 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral arterial disease; Platelet lysate
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet lysate (Active Comparator): A total of 5 ml platelet lysate will be intramuscularly injected in 4 doses with 2 week interval
  Interventions: Biological: Platelet lysate
- placebo (Placebo Comparator): A total of 5 ml of Normal Saline will be intramuscularly injected in 4 doses with 2 week interval
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Platelet lysate — Intramuscular injection of platelet lysate
  Arms: Platelet lysate
Biological: Placebo — intramuscular injection of normal saline
  Arms: placebo

SUMMARY:
Allogenic platelet lysate will be injected in the gastrocnemius of patients with peripheral arterial disease (PAD)

DETAILED DESCRIPTION:
Allogenic platelet rich plasma (PRP) will be collected from blood group AB donors. This plasma will be tested for the presence of any chronic infectious blood borne disease.

Platelet lysate will be then prepared from the tested PRP to be intramuscularly injected in patients with PAD

ELIGIBILITY:
Inclusion Criteria:

* Competent and willing to give informed consent, and to be available for all baseline treatment and follow up examinations required by the protocol.
* Gender: Male or female.
* Age group > 50 years.
* Established Critical limb ischemia (CLI), clinically and hemodynamically confirmed as per Rutherford 3, 4 and 5 with angiographic evidence of significant infra-inguinal arterial occlusive disease.
* History of intermittent claudication for > eight weeks.
* Limited exercise due to moderate to severe claudication.
* Resting ABI < 0.6, toe pressure ≤ 60 mm Hg, Toe Brachial index (TBI) <0.6, or TcPO2 ≤ 60 mmHg in the foot.
* Not eligible for surgical or radiological revascularization, and doesn't respond to best standard care delivered as confirmed by a vascular surgeon and/or physician.
* Fairly controlled diabetes (Hemoglobin A1c <10%).
* Normal liver enzymes, serum creatinine < 1.4
* Normal platelet count.
* On regular medication for hypertension if any.
* No evidence of malignancy
* Body mass index <30.

Exclusion Criteria:

* Women with child bearing potential, pregnant and lactating women.
* Rheumatoid Arthritis.
* History of neoplasm or malignancy in the past 10 years.
* Reported unstable cardiovascular disease, heart failure or symptomatic postural hypotension within 6 months before screening.
* Leg edema
* Inflammatory or progressive fibrotic disorder
* Renal insufficiency or failure
* History of infectious disorder (Human immunodeficiency virus (HIV) and/or hepatitis viruses).
* Chronic inflammatory disease
* History of stroke or myocardial infarction (< 3 months).
* Bleeding or clotting disorder, use of oral anticoagulant therapy (heparin, warfarin).

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 6 months
  Frequency and nature of adverse events occurring during a 6-month period following platelet lysate injection(s). This will be assessed by physical examination combined with a report with chemistry blood tests.

SECONDARY OUTCOMES:
Evaluation of the preliminary efficacy of the platelet lysate injection on patients' ABI | 12 months
  Positive changes in patients' Ankle brachial index (ABI)
Evaluation of the preliminary efficacy of the platelet lysate injection on patients' Toe pressure | 12 months
  Positive changes in patients' Toe pressure (mm Hg)
Evaluation of the preliminary efficacy of the platelet lysate injection on patients' TcPO2 | 12 months
  Positive changes in patients' Transcutaneous oxygen pressure (TcPO2)

CONTACTS AND LOCATIONS:
Overall Officials: Abdalla Awidi, MD, Study Director — Cell Therapy Center
Locations (1):
- Cell Therapy Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided